CLINICAL TRIAL: NCT01356251
Title: Mesothelioma From a Patient Perspective: A Survey of Psychosocial Needs and Exploration of Online Support for Patients
Brief Title: Psychosocial Needs and Exploration of Online Support for Patients With Mesothelioma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 11-066
Record Dates: First submitted 2011-05-17; First posted 2011-05-19 (Estimated); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Mesothelioma
Keywords: Quality of life; support group; questionnaires; Internet-based support group; 11-066
MeSH Terms: conditions — Mesothelioma | interventions — Surveys and Questionnaires

ARMS (2):
- Surgical group with mesothelioma (Experimental): The study proposed here has two parts: part 1 surveys mesothelioma patients' psychological and physical symptom burden and quality of life through a set of questionnaires that covers topics including coping, interpersonal support, mood, anxiety, and overall quality of life. In part 2, patients are invited to participate in an Internet-based discussion group.
  Interventions: Behavioral: Questionnaires & online virtual support group
- Non Surgical group with mesothelioma (Experimental): The study proposed here has two parts: part 1 surveys mesothelioma patients' psychological and physical symptom burden and quality of life through a set of questionnaires that covers topics including coping, interpersonal support, mood, anxiety, and overall quality of life. In part 2, patients are invited to participate in an Internet-based discussion group
  Interventions: Behavioral: Questionnaires & online virtual support group

INTERVENTIONS:
Behavioral: Questionnaires & online virtual support group — Part 1 surveys mesothelioma patients' psychological and physical symptom burden and quality of life by administering a set of questionnaires that covers topics including coping, interpersonal support, mood, anxiety, and overall quality of life. All mesothelioma patients who complete the questionnaires in part 1 will be offered an opportunity to participate in a trial of a therapeutic Internet-based discussion group. The groups will consist of either approximately 3-5 surgical patients or approximately 3-5 non-surgical patients. The groups will run for approximately 60 minutes once a week for six consecutive weeks.
  Arms: Surgical group with mesothelioma
Behavioral: Questionnaires & online virtual support group — Part 1 surveys mesothelioma patients' psychological and physical symptom burden and quality of life by administering a set of questionnaires that covers topics including coping, interpersonal support, mood, anxiety, and overall quality of life. All mesothelioma patients who complete the questionnaires in part 1 will be offered an opportunity to participate in a trial of a therapeutic Internet-based discussion group. The groups will consist of either 3-5 surgical patients or 3-5 non-surgical patients. The groups will run for approximately 60 minutes once a week for six consecutive weeks.
  Arms: Non Surgical group with mesothelioma

SUMMARY:
The aim of this study is to learn about how mesothelioma affects patients' emotional and physical well-being. Also, the investigators would like to learn more about what patients need and how they deal with this illness. This information can help us find ways to lessen physical and emotional strains. Part of the study tests an alternate way of giving emotional support through the Internet. By providing support online, patients can participate in the comfort of their home.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of pleural mesothelioma and receiving care at MSKCC
* At least 18 years of age or older
* Able to read and speak English
* Patients who choose to participate in the Internet-based discussion groups, need a telephone, a computer, Internet access, and an e-mail account.

Exclusion Criteria:

* Significant psychiatric or cognitive disturbance sufficient, in the investigator's judgment, to preclude providing informed consent or participating in a group-format intervention (i.e., acute psychiatric symptoms which require individual treatment).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2011-05 (Actual); Primary Completion 2023-02-06 (Actual); Study Completion 2023-02-06 (Actual)

PRIMARY OUTCOMES:
To describe the psychological needs of patients with mesothelioma. | 1 year
  Patients'psychological symptom burden will be assessed by the set of questionnaires administered in part 1 of the study. scores of the assessments of coping (28-item Brief Cope), social support (6-item SSQ-SF), depressive symptoms (20-item Zung), and quality of life (36-item FACT-Lung).

SECONDARY OUTCOMES:
the aim is to explore the acceptability and promise of an Internet-based discussion group for patients with mesothelioma. | 1 year
  The investigators will summarize acceptability and gather pilot data on the promise of the intervention. Acceptability in this study will be assessed through the enrollment rate (percentage of eligible individuals consented and recruited into the Internet-based discussion group). The adherence rate will be the percentage of enrolled patients who complete all virtual group sessions.

CONTACTS AND LOCATIONS:
Overall Officials: Christian Nelson, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm